CLINICAL TRIAL: NCT02799511
Title: Biomarkers for the Diagnosis of Transient Ischemic Attack
Acronym: MAESTRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-A00346-41
Record Dates: First submitted 2016-05-27; First posted 2016-06-15 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2019-12

CONDITIONS: Cerebrovascular Disorders; Ischemic Attack, Transient
Keywords: biological markers
MeSH Terms: conditions — Cerebrovascular Disorders; Ischemic Attack, Transient | interventions — Gene Expression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- protein expression (Other)
  Interventions: Biological: protein expression

INTERVENTIONS:
Biological: protein expression — Differential protein expression between the period of acute cerebral ischemia and the control period

SUMMARY:
A transient ischemic attack (TIA) should be considered an emergency prevention opportunity in order to avoid recurrence as cerebral infarction (CI) serious (fatal or disabling). Indeed, about 20% of patients who have IC had in previous days or weeks, a TIA, which can be defined as a brief episode of cerebral dysfunction (or eye) do not result in permanent brain damage and thus no sequelae. Moreover, about 20% of ischemic events observed in practice are AIT. Despite the progress achieved in the treatment in the acute phase of an IC, prevention remains the most effective way to fight against this disease. This prevention can be put in place before the occurrence of a first IC, or after a first IC, especially when minor as a TIA.

However, the diagnosis of TIA remains particularly difficult and it is necessary now to identify new tools for the diagnosis of transient ischemic attack. Our study focused on the identification of one or more molecules (called biological markers or biomarkers) present in the bloodstream of patients, which will serve to facilitate the differential diagnosis of patients with TIA.

ELIGIBILITY:
Inclusion Criteria:

* TIA lasting 18h
* NIHSS < 0
* MRI diffusion hypersignal less than 5 ml
* follow up during 3 month
* written informed consent prior to any study procedures

Exclusion Criteria:

* Pregnant or breastfeeding women
* major comorbidity (cancer, chronic infection)
* recent trauma (less than 30 days) (cranial or extracranial)
* Surgical or endovascular recent surgery(within 30 days).
* Any old brain injury
* Any acute pathology likely to induce inflammation, hemostasis disorders ...
* Contraindications to MRI: Patients with a pacemaker, an implanted material activated by an electrical, magnetic or mechanical carriers hemostatic clips intracerebral aneurysms or carotid arteries, bearing orthopedic implants, claustrophobic ...
* Patient under guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-03; Primary Completion 2019-01 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
change in proteomic analysis from MPs or from plasma. | baseline and 72h after TAI and 90 days after TAI
  Identify one or more markers of transient ischemic attack by a proteomic analysis from MPs or from plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- Caen University Hospital, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided